CLINICAL TRIAL: NCT06263790
Title: Intubating Laryngeal Mask vs Direct Laryngoscopy: a Crossover Randomized Controlled Preterm Manikin Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEOUNIPD1(2024)
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Neonatal Disease; Intubation; Difficult or Failed
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubation via laryngeal mask (Experimental): Participants will be required to position the endotracheal tube in the manikin via a laryngeal mask
  Interventions: Device: Intubating laryngeal mask
- Intubation via direct laryngoscope (Active Comparator): Participants will be required to position the endotracheal tube in the manikin via direct laryngoscopy
  Interventions: Device: Direct laryngoscopy

INTERVENTIONS:
Device: Intubating laryngeal mask — Intubation through a laryngeal mask
  Arms: Intubation via laryngeal mask
Device: Direct laryngoscopy — Intubation by using a direct laryngoscope
  Arms: Intubation via direct laryngoscope

SUMMARY:
The study aims to compare the success and time of intubation through an intubating laryngeal mask vs. direct laryngoscopy in a manikin simulating a term infant. In addition, we will assess the operator's opinion on the procedure.

This is an unblinded, randomized, controlled, crossover (AB/BA) pilot trial of intubation procedure through intubating laryngeal mask vs direct laryngoscopy in a manikin simulating a term newborn.

DETAILED DESCRIPTION:
Background: Endotracheal intubation is an important life-saving procedure for critically ill neonates. Furthermore, the procedure times are often longer than recommended by international guidelines, and repeated intubation attempts are associated with adverse events in unstable neonates.

Objectives: To compare success and time of intubation through intubating laryngeal mask vs. direct laryngoscopy in a manikin simulating a term infant. In addition, we will assess the operator's opinion on the procedure.

Methods: This is an unblinded, randomized, controlled, crossover (AB/BA) pilot trial of intubation procedure through intubating laryngeal mask vs direct laryngoscopy in a manikin simulating a term newborn. Participants will be level III NICU consultants and residents. Randomization will be performed using a computer-generated random assignment list. The primary outcome measure was the intubation success rate at the first attempt. Secondary outcome measures were the total time needed for the endotracheal tube positioning (calculated as the sum of the time of device positioning in all attempts), and the participant's opinion on using the device (evaluated using a Likert scale).

ELIGIBILITY:
Inclusion Criteria:

* Level III NICU consultants and residents will be eligible to participate in the study

Exclusion Criteria:

* None

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Success at the first attempt | 3 minutes after the initiation of the procedure
  The success of the first attempt will be defined as the achievement of the correct positioning of the endotracheal tube in the trachea as assessed by the external observer.

SECONDARY OUTCOMES:
Time of device positioning | 3 minutes after the initiation of the procedure
  Time of device positioning will be calculated as the sum of the time of device positioning in all attempts, as the procedure will be repeated in case of incorrect positioning
Participant's opinion on difficulty of the procedure | 5 minutes after end of the procedure
  Participants will report their opinion on insertion difficulty and overall difficulty using a Likert scale (1= not difficult, 5=very difficult)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madar J, Roehr CC, Ainsworth S, Ersdal H, Morley C, Rudiger M, Skare C, Szczapa T, Te Pas A, Trevisanuto D, Urlesberger B, Wilkinson D, Wyllie JP. European Resuscitation Council Guidelines 2021: Newborn resuscitation and support of transition of infants at birth. Resuscitation. 2021 Apr;161:291-326. doi: 10.1016/j.resuscitation.2021.02.014. Epub 2021 Mar 24. PMID 33773829
- [Background] Leone TA, Rich W, Finer NN. Neonatal intubation: success of pediatric trainees. J Pediatr. 2005 May;146(5):638-41. doi: 10.1016/j.jpeds.2005.01.029. PMID 15870667
- [Background] Sawyer T, Foglia E, Hatch LD, Moussa A, Ades A, Johnston L, Nishisaki A. Improving neonatal intubation safety: A journey of a thousand miles. J Neonatal Perinatal Med. 2017;10(2):125-131. doi: 10.3233/NPM-171686. PMID 28409758
- [Background] Gerstein NS, Braude DA, Hung O, Sanders JC, Murphy MF. The Fastrach Intubating Laryngeal Mask Airway: an overview and update. Can J Anaesth. 2010 Jun;57(6):588-601. doi: 10.1007/s12630-010-9272-x. Epub 2010 Jan 29. PMID 20112078
- [Background] Sauer CW, Kong JY, Vaucher YE, Finer N, Proudfoot JA, Boutin MA, Leone TA. Intubation Attempts Increase the Risk for Severe Intraventricular Hemorrhage in Preterm Infants-A Retrospective Cohort Study. J Pediatr. 2016 Oct;177:108-113. doi: 10.1016/j.jpeds.2016.06.051. Epub 2016 Jul 26. PMID 27470688
- [Derived] Monfredini C, Cavallin F, Ouedraogo P, Ezzahraoui L, Pasta E, Trevisanuto D, Villani PE. Intubating laryngeal airway vs. direct laryngoscope: a crossover randomized controlled neonatal manikin trial. Ital J Pediatr. 2025 Jun 20;51(1):196. doi: 10.1186/s13052-025-01988-8. PMID 40542416